CLINICAL TRIAL: NCT02484950
Title: A Prospective Randomized Trial of Biologic Augmentation With Mesenchymal Stem Cells in Patients Undergoing Arthroscopic Rotator Cuff Repair
Brief Title: Mesenchymal Stem Cell Augmentation in Patients Undergoing Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15042702
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Results first posted 2025-03-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: Mesenchymal stem cells

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotator cuff repair with stem cells (Experimental): Using clinically accepted methods, subjects will undergo bone marrow aspiration (from hip, proximal humerus or tibia) through a small incision prior to arthroscopy in the group undergoing MSC augmentation. They will then undergo arthroscopic full thickness rotator cuff repair using a double row, TOE anchor/suture technique with mesenchymal stem cell augmentation.
  Interventions: Biological: Mesenchymal stem cell augmentation in rotator cuff repair; Procedure: Standard arthroscopic rotator cuff repair
- Rotator cuff repair without stem cells (Placebo Comparator): Subjects will undergo arthroscopic full thickness rotator cuff repair using a double row, TOE anchor/suture technique, without augmentation of mesenchymal stem cells. To maintain patient blinding, all patients will receive a small incision around the site of expected bone marrow aspiration (hip, proximal humerus, or tibia), regardless of whether or not they receive bone marrow.
  Interventions: Procedure: Standard arthroscopic rotator cuff repair

INTERVENTIONS:
Biological: Mesenchymal stem cell augmentation in rotator cuff repair — Patients undergoing mesenchymal stem cell augmentation will receive a total injection of 6 milliliters (mL). Of this, 3 mL will be injected in the tendon at the junction between bone and tendon, while 3 mL will be injected in the bone at the site of the surgical footprint.
  Arms: Rotator cuff repair with stem cells
Procedure: Standard arthroscopic rotator cuff repair — All patients will undergo full thickness rotator cuff repair using a double row, transosseous-equivalent (TOE) repair with anchor/suture technique. Acromioplasty will be performed in all patients. Alternate procedures such as biceps tenotomy/tenodesis and distal clavicle excision will be performed at the discretion of the surgeon and recorded.

SUMMARY:
The primary objective of this study is to compare the clinical outcomes of arthroscopic rotator cuff repair with and without augmentation of mesenchymal stem cells (MSCs). Mesenchymal stem cells promote tissue regeneration by differentiating into adult cell lines and by supplying growth factors to their implanted environment. They have been shown to be effective in improving both overall healing and tendon integrity in rotator cuff repair. This study will follow 100 patients in the United States and track their clinical outcomes for at least one year post-operatively.

DETAILED DESCRIPTION:
Rotator cuff repair is one of the most commonly performed arthroscopic procedures in the United States, but re-tear remains a common long-term complication. This can lead to pain, decreased shoulder function, and the need for corrective surgery. Mesenchymal stem cells have been shown to improve healing rates in arthroscopic rotator cuff repair, primarily due to their retained ability to differentiate into several different adult cell lines, such as tenocytes, chondrocytes, and osteoblasts. MSCs further enhance the healing process by releasing growth factors into the local environment to promote tissue regeneration.

While MSC augmentation of arthroscopic rotator cuff repair has led to higher rates of healing and improved tendon integrity, there remains a paucity of data surrounding clinical improvement after the procedure. Outcomes such as post-operative strength, range of motion, and shoulder function have yet to be compared with standard rotator cuff repair. The incidence of post-operative persistent structural defects in the tendon after MSC augmentation must also be further elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patient is determined to have a full thickness rotator cuff tear (1-3 cm) or partial tear converted to a full-thickness tear-on the pre-operative MRI scan or found arthroscopically-and is scheduled to undergo surgical repair
* Written informed consent is obtained

Exclusion Criteria:

* Revision surgery
* Irreparable tear or partial repair
* Any patient lacking decisional capability
* Subscapularis involvement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil N Verma, MD, Principal Investigator — Midwest Orthopaedics at Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] MacDonald P, McRae S, Leiter J, Mascarenhas R, Lapner P. Arthroscopic rotator cuff repair with and without acromioplasty in the treatment of full-thickness rotator cuff tears: a multicenter, randomized controlled trial. J Bone Joint Surg Am. 2011 Nov 2;93(21):1953-60. doi: 10.2106/JBJS.K.00488. PMID 22048089
- [Background] Roy JS, MacDermid JC, Woodhouse LJ. Measuring shoulder function: a systematic review of four questionnaires. Arthritis Rheum. 2009 May 15;61(5):623-32. doi: 10.1002/art.24396. PMID 19405008
- [Background] Tashjian RZ, Deloach J, Green A, Porucznik CA, Powell AP. Minimal clinically important differences in ASES and simple shoulder test scores after nonoperative treatment of rotator cuff disease. J Bone Joint Surg Am. 2010 Feb;92(2):296-303. doi: 10.2106/JBJS.H.01296. PMID 20124055
- [Derived] Cole BJ, Kaiser JT, Wagner KR, Sivasundaram L, Otte RS, Tauro TM, White GM, Ralls ML, Yanke AB, Forsythe B, Romeo AA, Verma NN. Prospective Randomized Trial of Biologic Augmentation With Bone Marrow Aspirate Concentrate in Patients Undergoing Arthroscopic Rotator Cuff Repair. Am J Sports Med. 2023 Apr;51(5):1234-1242. doi: 10.1177/03635465231154601. Epub 2023 Feb 22. PMID 36811557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotator Cuff Repair With Stem Cells | Rotator Cuff Repair Without Stem Cells
Started | 28 | 34
Completed | 28 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rotator Cuff Repair With Stem Cells: Using clinically accepted methods, subjects will undergo bone marrow aspiration (from hip, proximal humerus or tibia) through a small incision prior to arthroscopy in the group undergoing MSC augmentation. They will then undergo arthroscopic full thickness rotator cuff repair using a double row, TOE anchor/suture technique with mesenchymal stem cell augmentation.
  Mesenchymal stem cell augmentation in rotator cuff repair: Patients undergoing mesenchymal stem cell augmentation will receive a total injection of 6 milliliters (mL). Of this, 3 mL will be injected in the tendon at the junction between bone and tendon, while 3 mL will be injected in the bone at the site of the surgical footprint.
  Standard arthroscopic rotator cuff repair: All patients will undergo full thickness rotator cuff repair using a double row, transosseous-equivalent (TOE) repair with anchor/suture technique. Acromioplasty will be performed in all patients. Alternate procedures such as biceps tenotomy/tenodesis and distal clavicle excision will be performed at the discretion of the surgeon and recorded.
  All patients underwent a shoulder exam pre-operatively as well as at 3 months, 6 months, 1 year and 2 years post-operatively. All patients completed the Standardized Shoulder Test (SST), ASES, Constant, SANE, and VR/SF-12 questionnaires preoperatively as well as 3 months, 6 months, 12 months, 18 months and 24 months postoperatively.
- Rotator Cuff Repair Without Stem Cells: Subjects will undergo arthroscopic full thickness rotator cuff repair using a double row, TOE anchor/suture technique, without augmentation of mesenchymal stem cells. To maintain patient blinding, all patients will receive a small incision around the site of expected bone marrow aspiration (hip, proximal humerus, or tibia), regardless of whether or not they receive bone marrow.
  Standard arthroscopic rotator cuff repair: All patients will undergo full thickness rotator cuff repair using a double row, transosseous-equivalent (TOE) repair with anchor/suture technique. Acromioplasty will be performed in all patients. Alternate procedures such as biceps tenotomy/tenodesis and distal clavicle excision will be performed at the discretion of the surgeon and recorded.
  All patients underwent a shoulder exam pre-operatively as well as at 3 months, 6 months, 1 year and 2 years post-operatively. All patients completed the Standardized Shoulder Test (SST), ASES, Constant, SANE, and VR/SF-12 questionnaires preoperatively as well as 3 months, 6 months, 12 months, 18 months and 24 months postoperatively.
- Total: Total of all reporting groups
Arm/Group | Rotator Cuff Repair With Stem Cells | Rotator Cuff Repair Without Stem Cells | Total
Number analyzed (Participants) | 28 | 34 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 8 | 14 | 22
Age, Continuous [Mean (Full Range); unit: years] | 49 [18 to 70] | 47 [18 to 70] | 48 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 8 | 14 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 20 | 25 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons (ASES) Score
Description: The American Shoulder and Elbow Surgeons (ASES) score is a patient-reported score that measures shoulder pain, activity level and stability.
  The score ranges from 0 to 100, with higher scores indicating better shoulder function.
  Excellent: 90-100 points Good: 70-89 points Fair: 40-49 points Poor: Less than 39 points
Time Frame: One year
Population: This study analyzed the efficacy of using autologous Bone Marrow Aspirate Concentrate (BMAC) compared with a control group in the recovery from rotator cuff surgery of the shoulder. The primary analysis focused on the American Shoulder and Elbow Surgeons (ASES) Score at 12 months post-surgery.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Rotator Cuff Repair With Stem Cells | Rotator Cuff Repair Without Stem Cells
Number analyzed (Participants) | 28 | 34
score on a scale | 87 [0 to 100] | 89 [0 to 100]

ADVERSE EVENTS:
Time Frame: 2 years
Description: There were no adverse events
Arm/Group | Rotator Cuff Repair With Stem Cells | Rotator Cuff Repair Without Stem Cells
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/34
Other Adverse Events (participants affected / at risk) | 0/28 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02484950/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02484950/ICF_002.pdf